CLINICAL TRIAL: NCT04456218
Title: Clinical Evaluation of a Custom-made and Disposable Endoscope System for Biliary Tract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chiao-Hsiung Chuang, Associate Professor, National Cheng-Kung University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: A-BR-108-097
Record Dates: First submitted 2020-06-14; First posted 2020-07-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Biliary Tract; Neoplasms; Stone - Biliary
MeSH Terms: conditions — Neoplasms; Cholecystolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biliary stone (Experimental): Participants who meet the criteria of biliary stone enrollment and are willing to join in this study will be applied to the custom-made endoscope system for biliary disease diagnosis.
  Interventions: Device: NCKU-scope-01 (a custom-made biliary endoscope system)
- Biliary stricture (Experimental): Participants who meet the criteria of biliary neoplasm enrollment and are willing to join in this study will be applied to the custom-made endoscope system for biliary disease diagnosis.
  Interventions: Device: NCKU-scope-01 (a custom-made biliary endoscope system)

INTERVENTIONS:
Device: NCKU-scope-01 (a custom-made biliary endoscope system) — The NCKU-scope-01 is a custom-made endoscope system for this study and it will be applied to help biliary disorders diagnosis

SUMMARY:
A disposable endoscopy system (NCKU-scope-01) was developed for the evaluation of bile duct stone or neoplasm. This system consists of a camera, light sources, a working channel, and a water injection channel. The endoscope could be inserted into the common bile duct via the working channel of a commercial duodenoscope. This study aims to test the feasibility and safety of this system. The efficacy of stone and neoplasm diagnosis will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complicated bile duct stone (stone size > 1.5 cm or number of stone > 3 )
* Patients with indeterminate biliary stricture or obstruction

Exclusion Criteria:

* Pregnant woman;
* Patients who are not suitable for ERCP (e.g. behavior disorder, major cognitive-perceptual deficit, etc.).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
A complete common bile duct accessing rate | 1 day
  To test the device's feasibility
Image quality evaluation: the light brightness and the imaging sharpness in Likert scale | 1 day
  To test the device's feasibility. About Likert scale, it range from 1 to 5 (1 is worse and 5 is better).

SECONDARY OUTCOMES:
Number of complications (ablation, bleeding, perforation in percentage) or system malfunction | 1 day
  To test the device's safety
In biliary stone arm: The biggest residual stone size (in cm). | 1 day
  The ability for residual stones diagnosis after initial ERCP stone extraction, compared with standard x-ray imaging)
In biliary stricture arm: Number of the lesions with or without presenting of the specific features for DDx of the benign or malignant stricture | 1 day
  The ability for differential diagnosis of benign or malignant stricture. The specific features include increased vascularity, irregular mucosa/nodularity, luminal narrowing, tumor vessel, mucosal lesion.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan